CLINICAL TRIAL: NCT02488902
Title: A Randomized, Double-blind, Placebo-controlled Evaluation of Increasing Doses of Weekly Tafenoquine for Chemosuppression of Plasmodium Falciparum in Semi-immune Adults Living in the Kassena-Nankana District of Northern Ghana
Brief Title: A Randomized, Double-blind, Placebo-controlled Evaluation of Increasing Doses of Weekly Tafenoquine for Chemosuppression of Plasmodium Falciparum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-8340
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — tafenoquine; Mefloquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Placebo
- Tafenoquine 25mg (Experimental): Tafenoquine was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Tafenoquine 25mg
- Tafenoquine 50mg (Experimental): Tafenoquine was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Tafenoquine 50mg
- Tafenoquine 100 mg (Experimental): Tafenoquine was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Tafenoquine 100 mg
- Tafenoquine 200 mg (Experimental): Tafenoquine was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Tafenoquine 200 mg
- Mefloquine 250 mg (Experimental): Mefloquine was administered initially as a loading course of one capsule daily for 3 days, followed by a weekly dosing regimen at the same dose.
  Interventions: Drug: Mefloquine 250 mg

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Tafenoquine 25mg — Tafenoquine 25mg
  Arms: Tafenoquine 25mg
Drug: Tafenoquine 50mg — Tafenoquine 50mg
  Arms: Tafenoquine 50mg
Drug: Tafenoquine 100 mg — Tafenoquine 100 mg
  Arms: Tafenoquine 100 mg
Drug: Tafenoquine 200 mg — Tafenoquine 200 mg
  Arms: Tafenoquine 200 mg
Drug: Mefloquine 250 mg — Mefloquine 250 mg
  Arms: Mefloquine 250 mg

SUMMARY:
This was a randomised, double-blind, placebo-controlled study to compare the efficacy of a range four weekly doses of tafenoquine, and weekly mefloquine, with placebo as chemosuppression of P. falciparum malaria. Medications and placebo were matched and a double-dummy technique enabled blinding of tafenoquine versus mefloquine.

ELIGIBILITY:
Inclusion Criteria:

* Willing subjects in good general health.

  * Males aged 18 to 60; females aged 50 to 60.
  * Subjects who planned to stay in the study area until the end of the study.

Exclusion Criteria:

* Subjects with any cardiovascular, liver, neurologic, or renal function abnormality which, in the opinion of the clinical investigators, would have placed them at increased risk of an adverse event or confused the result.

  * Subjects with a personal or family history of seizures or frank psychiatric disorder.
  * Females who had not ceased menstruation; a urine β-human chorionic gonadotrophin (β-HCG) test was to be performed at screening females who had ceased menstruation to exclude pregnancy as a cause.
  * Females who were lactating.
  * Subjects given antimalarial drugs for treatment within two weeks of study drug initiation.
  * Subjects with clinically significant abnormalities (to include but not limited to abnormal hepatic or renal function) as determined by history, physical and routine blood chemistry and haematology values.
  * Subjects with known hypersensitivity to any of the study drugs.
  * Subjects unwilling to remain in the area, report for drug administration or blood drawing during the 3-4 month duration of the study.
  * Subjects with G6PD deficiency (as determined by two separate qualitative tests per subject administered using distinct methods; methods used were visual dye and filter paper methods).
  * Subjects with any of the following laboratory values: haemoglobin (Hb) <8g/dL, platelets <80,000/mm3, white blood cell count (WBC) <3000/mm3, creatinine >1.5mg/dL, alanine transaminase (ALT) >60IU or 1+ haematuria as detected by urine dipstick.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 521 (Actual)
Dates: Start 1998-08; Primary Completion 1998-09 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
First occurrence of malaria infection | 16 weeks
  First occurrence of malaria infection as documented by a positive malaria smear.

SECONDARY OUTCOMES:
Time to confirmation of parasitaemia | 16 weeks
  Time to confirmation of parasitaemia as documented by two consecutive positive smears and the incidence density of parasitaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Braden Hale, MD, Principal Investigator — US Naval Medical Research Unit

REFERENCES:
- [Derived] Novitt-Moreno A, Ransom J, Dow G, Smith B, Read LT, Toovey S. Tafenoquine for malaria prophylaxis in adults: An integrated safety analysis. Travel Med Infect Dis. 2017 May-Jun;17:19-27. doi: 10.1016/j.tmaid.2017.05.008. Epub 2017 May 8. PMID 28495354